CLINICAL TRIAL: NCT01998789
Title: A Single Center, Open-label, Randomized, Controlled Pilot Trial to Evaluate the Efficacy and Safety of Everolimus Conversion Versus Standard Immunosuppression in Liver Transplant Recipients
Brief Title: Everolimus Post Orthotopic Liver Transplant
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tomoaki Kato (Other)
Responsible Party: Sponsor-Investigator, Tomoaki Kato, Chief, Division of Abdominal Organ Transplantation, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAL1602
Record Dates: First submitted 2013-11-25; First posted 2013-12-02 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Orthotopic Liver Transplant
Keywords: Liver Transplantation; Everolimus; Immunosuppression
MeSH Terms: interventions — Everolimus; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Everolimus Conversion Arm (Experimental): Everolimus will be initiated within 24 hours of baseline at a dose of 1 mg po BID (2 mg/day). Therapeutic Drug Monitoring will be performed throughout the study. Tacrolimus should be eliminated when the everolimus target range has been reached. Complete tacrolimus elimination will not occur earlier than 90 days post transplant and no later than 120 days post transplant. Enteric coated mycopenolic acid will be maintained for the duration of the study. Oral corticosteroids may not be eliminated sooner than 180 days post transplantation.
  Everolimus doses will be adjusted based on local lab results of everolimus trough levels.
  Interventions: Drug: Everolimus
- Standard Tacrolimus Immunosuppresion Arm (Active Comparator): Subjects will be maintained on standard maintenance immunosuppression per local protocol, consisting of a tacrolimus plus enteric coated mycophenolic acid. Oral corticosteroids may not be eliminated sooner than 180 days post transplantation.
  Tacrolimus doses will be adjusted based on local lab results of tacrolimus trough levels.
  Interventions: Drug: Standard Tacrolimus

INTERVENTIONS:
Drug: Everolimus — Everolimus will be initiated within 24 hours of baseline at a dose of 1 mg po BID (2 mg/day).
  Other Names: Zortress
  Arms: Everolimus Conversion Arm
Drug: Standard Tacrolimus — Subjects will be maintained on standard maintenance immunosuppression per local protocol, consisting of a tacrolimus plus enteric coated mycophenolic acid. Oral corticosteroids may not be eliminated sooner than 180 days post transplantation.
  Tacrolimus doses will be adjusted based on local lab results of tacrolimus trough levels.
  Other Names: Prograf
  Arms: Standard Tacrolimus Immunosuppresion Arm

SUMMARY:
The purpose of this study is to evaluate the efficacy of an everolimus conversion (EVR) protocol as compared to the standard tacrolimus (TAC) based protocol in liver transplant recipients, as determined by renal function, rejection rates, and progression to fibrosis (in HCV positive subjects). Additionally, safety profile and tolerability of these regimens will be assessed.

DETAILED DESCRIPTION:
The mainstay of maintenance immunosuppression post-transplantation includes a calcineurin inhibitor, either cyclosporine or tacrolimus. The introduction of calcineurin inhibitors led to a significant improvement in graft and patient outcomes post solid organ transplantation. However, one of the severe limitations of this class of drugs, is its associated nephrotoxicity. Data from the Scientific Registry of Transplant Recipients reveal that the incidence of stage 4 chronic kidney disease or stage 5 Chronic Kidney Disease (CKD) after Orthotopic Liver Transplantation (OLT) at 1, 3, and 5 years is 8%, 14%, and 18%, respectively, increasing to approximately 25% by 10 years after transplantation.Furthermore, renal dysfunction is associated with a four-fold increase in patient mortality post solid organ transplantation.

Several calcineurin inhibitor sparing and minimizing regimens have been studied. Most recently, in the phase III, randomized study in de novo liver transplant recipients,demonstrated significantly improved renal function in the tacrolimus minimization arm (everolimus plus tacrolimus one year post transplant.In fact superior renal function was achieved with the tacrolimus minimization arm one month after randomization and was maintained to Month 12. With this pilot study, we aim to compare the efficacy of the standard immunosupression post liver transplant with Tacrolimus and Mycophenolic acid (Myfortic)with calcineurin sparing regimen using the combination of everolimus and enteric coated mycophenolic acid, as determined by the estimated Glomerular filtration rate (GFR) at one year post transplant, with acceptable rates of biopsy proven rejection.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide informed consent and adhere to study regimen
* Recipients of primary liver transplant from deceased or living donor
* 18 years of age or greater
* Lab Model For End-Stage Liver Disease (MELD) score ≤ 30
* Abbreviated Modification of Diet in Renal Disease (MDRD) eGFR ≥ 30 mL/min/1.73

Key Exclusion Criteria:

* Recipient of multiple solid or organ transplant, or have previously received and organ transplant
* Women of child-bearing potential unless they are willing to participate in adequate contraception methods as outlined in the study.
* HIV infection (results obtained 6 months prior to screening is acceptable)

Key Exclusion-Baseline/ Randamization

* Severe hypercholesterolemia (> 350 mg/dL) or hypertriglyceridemia (> 500 mg/dL) within 30 days prior to baseline.
* Thrombocytopenia (platelets < 50,000/mm3)
* Absolute neutrophil count of < 1000/mm3 or white blood cell count of < 2000/mm3
* Subjects in a critical care unit requiring life support measures such as mechanical ventilation, dialysis, requirement of vasopressor agents
* Liver allograft is functioning at an unacceptable level as defined by the Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Total Bilirubin levels > 3 times upper limit of normal (ULN) and Alkaline Phosphatase (AlkP) and Gamma-glutamyltransferase (GGT) levels > 5 times ULN
* Diagnosis of autoimmune hepatitis, primary biliary cirrhosis and primary sclerosing cholangitis
* Hepatocellular carcinoma with evidence of macrovascular invasion on explanted liver or evidence of extrahepatic spread
* Inability to take medications by mouth
* Renal insufficiency, as defined by abbreviated MDRD eGFR < 30 mL/min/1.73m2, or requirement of dialysis, that does not recover prior to baseline
* Episode of acute rejection requiring antibody therapy or more than one steroid treated episode of acute rejection
* Subjects with a confirmed spot urine protein/creatinine ratio that indicates ≥1g/24h of proteinuria.
* Subtherapeutic trough levels of tacrolimus during the week prior to baseline (subject must have at least one tacrolimus level ≥ 8 ng/mL)
* The presence of thrombosis via Doppler ultrasound of the major hepatic arteries, major hepatic veins, portal vein and inferior vena cava.
* Presence of clinically significant wound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-10; Primary Completion 2018-06 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Change in estimated Glomerular Filtration Rate (eGFR) | Baseline and 12 months post transplant
  Comparison of change in Renal function, as measured by eGFR from baseline to 12 months post liver transplantation, in subjects maintained on an everolimus conversion regimen versus those maintained on a standard tacrolimus based regimen.

SECONDARY OUTCOMES:
Change in estimated Glomerular Filtration Rate (eGFR) | Baseline and 24 months post liver transplantation
  1. Comparison of renal function, as measured eGFR from baseline to 24 months post liver transplantation, in subjects maintained on an everolimus conversion regimen versus those maintained on a standard tacrolimus based regimen.
  2. To compare the incidence of renal insufficiency, defined as GFR<30 or need for dialysis at 12 months and 24 months post liver transplantation, in subjects maintained on an everolimus conversion regimen versus those maintained on a standard tacrolimus based regimen.
Proportion of HCV patients who develop stage 2 of 4 or greater fibrosis, liver failure, or fibrosing cholestatic hepatitis (FCH) at month 12 and 24 | Up to 24 months post liver transplantation
  To determine whether everolimus conversion post liver transplantation reduces progression of fibrosis at 12 and 24 months post transplant as compared to standard tacrolimus based immunosuppression in liver transplant recipients with Hepatitis C as measured by:
  Proportion of patients who develop stage 2 of 4 or greater fibrosis, liver failure, or fibrosing cholestatic hepatitis (FCH) at month 12 and 24
Composite Efficacy Failure Rate | Up to 24 months
  To compare the composite efficacy failure rates of treated biopsy proven acute rejection, graft loss, death, or loss to follow up with Everolimus conversion arm to standard immunosuppression with Tacrolimus based arm at 12 and 24 months after liver transplant.
  To compare each component of the composite efficacy failure rates between Everolimus conversion and standard Tacrolimus arm.
  To compare the composite graft failure or death or loss of follow up between the two arms.
  To Evaluate acute rejection by incidence, time to interval and severity.
Incidence of Hepatocellular Carcinoma (HCC) Recurrence | Up to 12 months post transplant
  In subjects with Hepatocellular carcinoma (HCC), to compare the incidence of HCC recurrence at 12 months post transplantation between the Everolimus conversion arm and the standard tacrolimus based arm, as evaluated by radiological studies, biopsy findings, and/or AFP levels.

CONTACTS AND LOCATIONS:
Overall Officials: Tomoaki Kato, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center-NYPH, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided